CLINICAL TRIAL: NCT07141238
Title: Analysis of Microplastics in Pediatric Inflammatory Bowel Disease Using Raman Spectroscopy: A Multi-Matrix Study
Brief Title: Microplastic Analysis in Pediatric Inflammatory Bowel Disease
Acronym: MAP-IBD
Status: Recruiting | Type: Observational
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Sponsor
Other Study IDs: MAP-IBD-2025
Record Dates: First submitted 2025-08-18; First posted 2025-08-26 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Crohn Disease; Pediatric Inflammatory Bowel Diseases; Ulcerative Colitis (UC); Inflammatory Bowel Disease (IBD)
Keywords: Microplastics; Pediatric Inflammatory Bowel Disease; Raman Spectroscopy; Environmental exposure; Ulcerative Colitis; Crohn's Disease
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Intestinal tissue biopsies, stool samples, urine samples, blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pediatric IBD group: Children diagnosed with inflammatory bowel disease (Crohn's disease or ulcerative colitis) undergoing clinically indicated endoscopy. Biological samples, including intestinal biopsies, stool, urine, and blood, will be collected and analyzed for microplastic content using Raman spectroscopy.
  Interventions: Other: Environmental microplastic exposure
- Control group: Children without a diagnosis of IBD undergoing endoscopy for non-inflammatory indications (e.g., polyps, anemia). Biological samples, including intestinal biopsies, stool, urine, and blood, will be collected and analyzed for microplastic content using Raman spectroscopy.
  Interventions: Other: Environmental microplastic exposure

INTERVENTIONS:
Other: Environmental microplastic exposure — Exposure to environmental microplastics measured by their presence in intestinal tissue, blood, urine, and stool using Raman spectroscopy. This study does not assign any exposure or treatment; it investigates the existing presence of microplastics as an environmental factor of interest.

SUMMARY:
The goal of this observational study is to measure and compare the presence of microplastics in children with inflammatory bowel disease (IBD) and children without IBD. The main questions it aims to answer are:

Are microplastics detectable in different biological samples from children? Are there differences in microplastic burden between children with and without IBD?

Researchers will collect biological samples including: intestinal tissue (from routine endoscopy), stool, urine, blood.

Raman spectroscopy will be used to detect and characterize microplastics in each sample type. Participants will not receive any medication or intervention as part of this study. All samples will be collected during standard clinical procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age <18 years
* Undergoing clinically indicated gastrointestinal endoscopy
* For IBD group: confirmed diagnosis of Crohn's disease or ulcerative colitis
* For control group: no current or past diagnosis of IBD

Exclusion Criteria:

* Age 18 years or older
* Lack of informed consent from legal guardian
* Lack of written assent from the participant if age ≥13 years

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients undergoing endoscopy at a tertiary care academic hospital. The study includes children with confirmed inflammatory bowel disease and children undergoing endoscopy for other indications as controls.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-06-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Presence and concentration of microplastics in intestinal tissue samples | Day of endoscopy (Baseline)
  Quantification of microplastics (number of particles per gram of tissue) detected using Raman spectroscopy in intestinal mucosal biopsies collected during clinically indicated endoscopy.

SECONDARY OUTCOMES:
Comparison of microplastic burden between children with IBD and controls | Baseline (Day of sample collection)
  Assessment of differences in all biological matrices (tissue, stool, blood, urine) between children with inflammatory bowel disease and controls

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Gdańsk, Department of Pediatrics, Gastroenterology, Allergolgy and Nutrition, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: No